CLINICAL TRIAL: NCT01188473
Title: Safety and Efficacy of Early Initiation of Noninvasive Positive Pressure Ventilation in Pediatric Patients Admitted With Status Asthmaticus
Brief Title: Early Noninvasive Positive Pressure Ventilation in Children With Status Asthmaticus
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Pilot early noninvasive ventilation on all children who met the criteria was effective.
Sponsor: Southern Illinois University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAS-SIU-10-005
Record Dates: First submitted 2010-08-23; First posted 2010-08-25 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Status Asthmaticus
Keywords: Status Asthmaticus; Noninvasive Positive Pressure Ventilation; Asthma in Children
MeSH Terms: conditions — Status Asthmaticus | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NPPV plus standard of care (Experimental): NPPV initiated early and for a prolonged period of time in addition to standard of care in the management of children admitted to the hospital with status asthmaticus
  Interventions: Other: NPPV plus standard of care
- Control: standard of care alone (No Intervention): standard of care in the management of children admitted to the hospital with status asthmaticus

INTERVENTIONS:
Other: NPPV plus standard of care — Patients in the NPPV group were fitted with a nasal mask with gel seals (Comfortgel Masks, Respironics) and placed on the BiPAP Machine (Vision Bipap, Respironics). To optimize patient cooperation, the mask was initially applied manually to the patient's face. After a short adaptation period, it was firmly applied on the face by head straps to minimize air leak without causing skin injury. Pressures were initially set low for comfort and acceptance while being placed on the machine. The inspiratory positive airway pressure (IPAP) was gradually increased to 8 cm H2O in order to achieve a tidal volume of 6-9 ml/kg and the end expiratory positive airway pressure (EPAP) to 5 cm H 2O. These settings remained unchanged throughout the study period.
  Other Names: Comfortgel Masks, Respironics; Vision Bipap, Respironics
  Arms: NPPV plus standard of care

SUMMARY:
Status asthmaticus is recognized as a common cause of morbidity in children in the United States. In recent years, hospitalization rates have reached an all time high. This study will evaluate the safety, tolerability and clinical benefit of adding Noninvasive Positive Pressure Ventilation (NPPV)to regular care in children with moderate to moderately severe status asthmaticus.

DETAILED DESCRIPTION:
Status asthmaticus is defined as severe asthma that fails to respond to inhaled short acting β agonists (SABA), oral or intravenous steroids, and oxygen, leading to hospital admission for further management (1). In 2004, asthma exacerbations led to 3% (198,000) of all hospitalizations and 2.5 deaths per 1 million populations in the 0-17 year age group (2).

This prospective, unblinded, randomized controlled, pilot clinical trial will compare NPPV plus standard of care versus standard of care alone in children admitted for status asthmaticus. NPPV refers to the delivery of pressurized gas through an external interface such as a nasal or oronasal mask, connected to a pressure targeted ventilator. In other words, it provides ventilator support without the use of an endotracheal tube.

This study will investigate the safety, tolerability and efficacy of early initiation of non-invasive NPPV in pediatric patients admitted with status asthmaticus.

ELIGIBILITY:
Inclusion Criteria:

* children, 1- 18 years of age, with a known history of asthma admitted to the PICU at St John's Children's Hospital with status asthmaticus
* clinical asthma score (CAS) between 3 - 8 after receiving one dose of systemic steroid, 1 hour of continuous albuterol (SABA), and 3 doses of ipratropium bromide
* written informed consent from the patient's parent or legal guardian

Exclusion Criteria:

* no previous history of asthma,
* absence of airway protective reflexes,
* absence of respiratory drive,
* excessive oral secretions,
* need for emergent intubation as determined by the attending physician,
* facial or airway anomaly or injury precluding the use of tight fitting mask

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
clinical asthma score (CAS) | initiation, 2 hours, 4-8 hours, 12-16 hours and 24 hours after initiation
  clinical evaluations such as wheezing, degree of air exchange, respiratory rate, I&E ratio, retractions

SECONDARY OUTCOMES:
heart rate | initiation, 2 hours, 4-8 hours, 12-16 hours and 24 hours after initiation
  determined by heart monitor
being able to wear the mask | initiation, 2 hours, 4-8 hours, 12-16 hours and 24 hours after initiation
  Patient is able to keep the mask on for 24 hours.
transcutaneous oxygen saturation | initiation, 2 hours, 4-8 hours, 12-16 hours and 24 hours after initiation
mental status | initiation, 2 hours, 4-8 hours, 12-16 hours and 24 hours after initiation
  observation of activity level, agitation, etc.
supplemental oxygen | initiation, 2 hours, 4-8 hours, 12-16 hours and 24 hours after initiation
NPPV related side effects | initiation, 2 hours, 4-8 hours, 12-16 hours and 24 hours after initiation
  NPPV related side effects could be minor including nasal bridge pain and skin irritation, gastric insufflations, sinus and ear pain, and dry eyes

CONTACTS AND LOCATIONS:
Overall Officials: Sangita Basnet, MD, Principal Investigator — Southern Illinois University School of Medicine
Locations (1):
- Southern Illinois University School of Medicine, Springfield, Illinois, United States